CLINICAL TRIAL: NCT02708030
Title: Efficacy of Ketogenic Diet, Modified Atkins Diet and Low Glycemic Index Therapy Diet Among Children With Drug Resistant Epilepsy: A Randomised Non-Inferiority Trial
Brief Title: Dietary Therapy In Epilepsy Treatment (DIET-Trial): A Randomised Non Inferiority Trial Comparing KD, MAD & LGIT for Drug Resistant Epilepsy
Acronym: DIET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD Vs MAD Vs LGIT
Record Dates: First submitted 2016-02-22; First posted 2016-03-15 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Diet, Ketogenic; mycophenolic adenine dinucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketogenic Diet (Active Comparator): Ketogenic diet (KD) will be administered by the non-fasting protocol. The child will be admitted to the hospital, and KD will be started in 1:1 ratio. The ratio will increased every 48hours to a maximum of 4:1 or ketosis (urinary ketones 40-80mg/dL) is attained. The child will thereafter be discharged and followed up on Out patient basis.
  Interventions: Other: Ketogenic Diet
- Modified Atkins Diet (Experimental): Modified Atkins Diet (MAD) will be administered on out patient basis. Parents of children will be advised to monitor for seizure frequency and ketosis at home.
  Interventions: Other: MAD
- Low Glycemic Index Therapy (Experimental): Low Glycemic Index Therapy (LGIT) will be administered on out patient basis. Parents of children will be advised to monitor for seizure frequency and ketosis at home.
  Interventions: Other: LGIT

INTERVENTIONS:
Other: Ketogenic Diet — The children with the drug resistant epilepsy will go through a run in period of 4 weeks during which each child will undergo a detailed detailed clinical evaluation according to a structured proforma, and baseline investigations. The patients in KD arm will be admitted to the hospital for initiation of diet.
  Arms: Ketogenic Diet
Other: MAD — The children with the drug resistant epilepsy will go through a run in period of 4 weeks during which each child will undergo a detailed detailed clinical evaluation according to a structured proforma, and baseline investigations. Following the run in period of 4 weeks, the patients will be randomized to the MAD or LGIT or KD arm. MAD will be initiated on out patient basis.
  Arms: Modified Atkins Diet
Other: LGIT — The children with the drug resistant epilepsy will go through a run in period of 4 weeks during which each child will undergo a detailed detailed clinical evaluation according to a structured proforma, and baseline investigations. Following the run in period of 4 weeks, the patients will be randomized to the MAD or LGIT or KD arm. LGIT will be initiated on out patient basis.
  Arms: Low Glycemic Index Therapy

SUMMARY:
This randomised trial is undertaken to assess whether MAD or LGIT is non-inferior to KD with regard to seizure control at twenty-four weeks among children with drug resistant epilepsy. The hypothesis of the study is that in 1 to 15-year-old children with drug resistant epilepsy, use of Modified Atkins Diet (MAD) or Low Glycemic Index Therapy (LGIT) as an add on to the ongoing anti-epileptic drugs would not be inferior to ketogenic diet by >15% in terms of seizure reduction from baseline seizure frequency at 24 weeks.

The primary outcome of the study is to determine the efficacy of MAD as compared to KD and LGIT as compared to KD for seizure reduction in drug resistant epilepsy following 24 weeks of dietary therapy in 1 to 15-year-old children on anti-epileptic drugs. The change in seizure frequency will be estimated as percentage change in seizure reduction at 24 weeks as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1-15 years with drug resistant epilepsy (Drug resistant epilepsy for the study will be defined as seizure frequency >4 seizures per month, and treatment failure of ≥2 prescribed antiepileptic drugs).
2. Willing to come for regular follow up

Exclusion Criteria:

1. Surgically remediable cause for drug resistant epilepsy
2. Proven inborn error of metabolism except those in which KD is indicated (i.e., Pyruvate Carboxylase deficiency and GLUT-1 Deficiency)
3. Previously received KD, MAD or LGIT
4. Known case of

   1. Chronic kidney disease
   2. Chronic liver disease/ GI illness
   3. Chronic heart disease (congenital and acquired)
   4. Chronic respiratory illness

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Percentage change in seizure frequency after 24 weeks of dietary therapy as compared to baseline, in the arm KD as compared to MAD and in the arm KD as compared to LGIT | Baseline and six months
  Percentage change in seizure frequency will be estimated as mean number of weekly seizures over preceding 4 weeks after 24 weeks of dietary therapy divided by mean number of weekly seizures over preceding 4 weeks at the baseline.
  It will be calculated for each of the three arms (KD; MAD; LGIT) and KD will compared to MAD and LGIT individually as the primary outcome.

SECONDARY OUTCOMES:
Percentage change in seizure frequency after 24 weeks of dietary therapy as compared to baseline, in the arm MAD as compared to LGIT | Baseline and twenty-four weeks
  Percentage change in seizure frequency will be estimated as mean number of weekly seizures over preceding 4 weeks after 24 weeks of dietary therapy divided by mean number of weekly seizures over preceding 4 weeks at the baseline. Change in seizure frequency in MAD and LGIT arm will be compared
Proportion of patients who achieve >50% seizure reduction from baseline at 24 weeks after diet initiation | Baseline and twenty-four weeks
  Proportion of patients who achieve >50% seizure reduction from baseline at 24 weeks after diet initiation
Estimate behavior change as measured by Childhood behavior checklist in each of three arms at baseline, 12 weeks and 24 weeks after dietary therapy | Baseline, twelve weeks, and twenty-four weeks
Estimate cognition change as assessed by Vineland Social Maturity Scale in each of three arms at baseline, 12 weeks and 24 weeks after dietary therapy | Baseline and twenty-four weeks
Evaluate GI adverse events (diarrhoea, constipation and vomiting) assessed by parental questionnaire in each of the three arms at baseline and six months after therapy | Baseline and twenty-four weeks
Evaluate change in serum levels of micronutrients by laboratory testing in each of three arms at baseline and six months after therapy | Baseline and twenty-four weeks
  Micronutrients like copper, zinc, retinol and vitamin E would be compared
Evaluate omega3 polyunsaturated fatty acid levels and correlate it with change in seizure frequency | Baseline and twenty-four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sondhi V, Agarwala A, Pandey RM, Chakrabarty B, Jauhari P, Lodha R, Toteja GS, Sharma S, Paul VK, Kossoff E, Gulati S. Efficacy of Ketogenic Diet, Modified Atkins Diet, and Low Glycemic Index Therapy Diet Among Children With Drug-Resistant Epilepsy: A Randomized Clinical Trial. JAMA Pediatr. 2020 Oct 1;174(10):944-951. doi: 10.1001/jamapediatrics.2020.2282. PMID 32761191
- [Derived] Martin-McGill KJ, Bresnahan R, Levy RG, Cooper PN. Ketogenic diets for drug-resistant epilepsy. Cochrane Database Syst Rev. 2020 Jun 24;6(6):CD001903. doi: 10.1002/14651858.CD001903.pub5. PMID 32588435